CLINICAL TRIAL: NCT04746365
Title: Ivermectin Role in Severe Covid-19 Treatment; a Double-blinded, Randomized Clinical Trial
Brief Title: Ivermectin Role in Covid-19 Clinical Trial
Acronym: IRICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elaraby Hospital (Other)
Collaborators: Shebin El-Kom Teaching Hospital (Other)
Responsible Party: Principal Investigator, Hozaifa Elsawah, Clinical Pharmacist, Elaraby Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1029076; 2101001 (Registry Identifier: IRICT trial)
Record Dates: First submitted 2021-02-06; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, controlled clinical trial
Who Masked: Participant, Care Provider
Masking Description: Unlabelled tablets were prepared for each patient in a special envelope in a time-based manner in the central pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ivermectin (Experimental): ivermectin was given as a total daily dose of 36 mg on days 0, 3, 6. The daily dose was divided into 3 equal doses of 12 mg (2 tablets) every 8 hours
  Interventions: Drug: ivermectin
- hydroxychloroquine (Experimental): hydroxychloroquine was given as 200 mg (one tablet) every 12 hours for 5 days
  Interventions: Drug: hydroxychloroquine
- Placebo (Placebo Comparator): Unlabelled standard treatment according to the clinical condition of patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ivermectin — ivermectin is anthelmintic
  Arms: ivermectin
Drug: hydroxychloroquine — hydroxychloroquine is antimalarial.
  Arms: hydroxychloroquine
Drug: Placebo — Standard treatments
  Arms: Placebo

SUMMARY:
Because ivermectin is being used to treat COVID-19 with insufficient evidence, the investigator conducted a randomized clinical trial to investigate the efficacy and safety of ivermectin in comparison to hydroxychloroquine and placebo in severe COVID-19 patients. The study was conducted in Shebin-Elkom teaching hospital and recruited patients from December 6, 2020, to January 31, 2021.

DETAILED DESCRIPTION:
This study is an adaptive, randomized, double-blinded, controlled trial to evaluate the safety and efficacy of therapeutic agents in hospitalized adult patients diagnosed with COVID-19. The study is a single-center trial that will be conducted in Shebin Elkom teaching hospital. The study will be a series of 3-arm comparisons between two different investigational therapeutic agents (Ivermectin and Hydroxychloroquine) and a placebo. There will be interim monitoring to allow early stopping for futility, efficacy, or safety. Because of the possibility that background standards of supportive care may evolve/improve over time as more is learned about the successful management of COVID-19, comparisons of safety and efficacy will be based on data from concurrently randomized participants. An independent data and safety monitoring board (DSMB) will actively monitor interim data to make recommendations about early study closure or changes to study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
2. Understands and agrees to comply with planned study procedures.
3. Agrees to the collection of OP swabs and venous blood per protocol.
4. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other
6. Severe cases according to WHO definition.

Exclusion Criteria:

1. ALT/AST > 5 times the upper limit of normal.
2. Mortality within 12 hours of admission.
3. Pregnancy.
4. Anticipated transfer to another hospital within 24 hours.
5. Allergy to any study medication commercial or public health assay in any specimen prior to randomization.
6. Mechanically ventilated on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Reduction in the WHO ordinal scale of clinical status by at least two points | 14 days
  The ordinal scale consists of 7 points, the maximum score is 7 which indicates a worst outcome, while the minimum score is 1 which indicates a better outcome
Time to discharge | within 14 days
  time to discharge to home after no more need for hospitalization

SECONDARY OUTCOMES:
Mortality | 14 days
  All-causes mortality

OTHER OUTCOMES:
Adverse events | 14 days
  Grade 3 and 4 adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shebin-Elkom teaching hospital, Shibīn al Kawm, Menoufia, Egypt

REFERENCES:
- [Derived] Elshafie AH, Elsawah HK, Hammad M, Sweed EM, Seif AS, Abdel Ghaffar MM, Goda FM, Mosalam EM, Abdallah MS. Ivermectin role in COVID-19 treatment (IRICT): single-center, adaptive, randomized, double-blind, placebo-controlled, clinical trial. Expert Rev Anti Infect Ther. 2022 Oct;20(10):1341-1350. doi: 10.1080/14787210.2022.2098113. Epub 2022 Jul 12. PMID 35788169